CLINICAL TRIAL: NCT00916006
Title: A Multi-center, Randomized, Parallel Group, Double-blind, Vehicle-controlled Study to Evaluate the Efficacy and Safety of PEP005 (Ingenol Mebutate) Gel, 0.015% In Patients With Actinic Keratoses ON the Head (Face or Scalp) (REGION-IIa)
Brief Title: A Multi-center Study to Evaluate the Efficacy and Safety of PEP005 (Ingenol Mebutate) Gel, When Used to Treat Actinic Keratoses on the Head (Face or Scalp)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Peplin (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PEP005-016
Record Dates: First submitted 2009-06-04; First posted 2009-06-08 (Estimated); Results first posted 2012-03-21 (Estimated); Last update posted 2015-04-02 (Estimated); Status verified 2015-03

CONDITIONS: Actinic Keratosis
Keywords: Peplin; Actinic keratosis; PEP005
MeSH Terms: conditions — Keratosis, Actinic | interventions — 3-ingenyl angelate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PEP005 gel (Experimental): PEP005 gel, 0.015% applied once daily for three consecutive days
  Interventions: Drug: PEP005 Gel
- Vehicle gel (Placebo Comparator): Vehicle gel applied once daily for three consecutive days
  Interventions: Drug: Vehicle gel

INTERVENTIONS:
Drug: PEP005 Gel — 0.015%, three day treatment
  Other Names: PEP005
  Arms: PEP005 gel
Drug: Vehicle gel — Vehicle gel, three day treatment
  Other Names: Placebo
  Arms: Vehicle gel

SUMMARY:
This Phase III study is designed to assess the efficacy and safety of PEP005 Gel, 0.015% when applied to an area of skin containing 4-8 AK lesions on the face or scalp.

ELIGIBILITY:
Inclusion Criteria:

* Patient is male or female and at least 18 years of age
* Female patients must be of either:

  * Non-childbearing potential, post-menopausal
  * Childbearing potential, provided there are negative serum and urine pregnancy test results prior to study treatment, to rule out pregnancy

Exclusion Criteria:

* Cosmetic or therapeutic procedures within 2 weeks and 2cm of the selected treatment area
* Treatment with immunomodulators, or interferon/ interferon inducers or systemic medications that suppress the immune system within 4 weeks
* Treatment with 5-FU, imiquimod, diclofenac, or photodynamic therapy: within 8 weeks and 2 cm of the selected treatment area

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 269 (Actual)
Dates: Start 2009-06; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Bauer, MD, Study Director — Chief Medical Officer
Locations (21):
- United States (19):
  - Dermatology Research Associates, Los Angeles, California
  - Dermatology Specialists Inc, Oceanside, California
  - Skin Surgery Medical Group Inc., San Diego, California
  - Conant Medical Group, San Francisco, California
  - University of Miami, Skin Research Camp, Miami, Florida
  - Atlanta Dermatology, Vein & Research Center, LLC, Alpharetta, Georgia
  - Medaphase Inc, Newnan, Georgia
  - Glazer Dermatology, Buffalo Grove, Illinois
  - Dawes Fretein Clinical Research Group, LLC, Indianapolis, Indiana
  - Pedia Research LLC, Owensboro, Kentucky
  - Hamzavi Dermatology, Fort Gratiot, Michigan
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Wake Research Associates, Raleigh, North Carolina
  - Dermatology Research Associates, Nashville, Tennessee
  - J & S Studies, Inc., College Station, Texas
  - Dermatology Associates of Tyler, Tyler, Texas
  - Center for Clinical Studies, Webster, Texas
  - Dermatology Research Center, Inc., Salt Lake City, Utah
  - Virginia Clinical Research, Inc, Norfolk, Virginia
- Australia (2):
  - Southderm Pty Ltd, Kogarah, New South Wales
  - St George Dematology and Skin Cancer Centre, Kogarah, New South Wales

REFERENCES:
- [Derived] Lebwohl M, Swanson N, Anderson LL, Melgaard A, Xu Z, Berman B. Ingenol mebutate gel for actinic keratosis. N Engl J Med. 2012 Mar 15;366(11):1010-9. doi: 10.1056/NEJMoa1111170. PMID 22417254
- See also: Food and Drug Authority — http://www.fda.gov
- See also: Therapeutic Goods Administration — http://www.tga.gov.au

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study PEP005-016 was conducted at 21 study centers in the United States and Australia. A total of 269 patients were randomized. Patient screening was started on 01 June 2009. The first patient was randomized on 05 June 2009 and the last patient completed the Day 57 visit on 10 September 2009
Groups:
- PEP005 (Ingenol Mebutate) Gel, 0.015%: PEP005 (ingenol mebutate) Gel 0.05% once daily for 3 consecutive days
- Vehicle: Vehicle gel once daily for 3 consecutive days
Period: Overall Study
Arm/Group | PEP005 (Ingenol Mebutate) Gel, 0.015% | Vehicle
Started | 135 | 134
Completed | 132 | 127
Not Completed | 3 | 7
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 2 | 5
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PEP005 (Ingenol Mebutate) Gel, 0.015% | Vehicle | Total
Number analyzed (Participants) | 135 | 134 | 269
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 71 | 77 | 148
  >=65 years | 64 | 57 | 121
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 14 | 33
  Male | 116 | 120 | 236
Region of Enrollment [Number; unit: participants]
  United States | 125 | 126 | 251
  Australia | 10 | 8 | 18

OUTCOME MEASURES:

1. Primary Outcome: Patients With Complete Clearance of Actinic Keratosis (AK) Lesions.
Description: Complete clearance rate of actinic keratosis (AK) lesions, defined as the proportion of patients with no clinically visible AK lesions in the selected treatment area.
Time Frame: 57 days
Population: Intention to treat population
Measure: Number; unit: participants
Groups:
- PEP005 (Ingenol Mebutate) Gel: PEP005 (ingenol mebutate) Gel 0.05% once daily for 3 consecutive days
- Vehicle Gel: Vehicle Gel once daily for 3 consecutive days
Arm/Group | PEP005 (Ingenol Mebutate) Gel | Vehicle Gel
Number analyzed (Participants) | 135 | 134
participants | 50 | 3
Statistical Analysis 1: Comparison: PEP005 (Ingenol Mebutate) Gel vs Vehicle Gel; Test type: Superiority or Other; p = 0.001, Cochran-Mantel-Haenszel

2. Secondary Outcome: Patients With Partial Clearance of Actinic Keratosis (AK)
Description: Patients with partial clearance defined as ≥ 75% reduction in the number of actinic keratosis (AK) lesions identified at baseline in the treatment area
Time Frame: baseline and 57 days
Population: Intention to treat population
Measure: Number; unit: participants
Arm/Group | PEP005 (Ingenol Mebutate) Gel | Vehicle Gel
Number analyzed (Participants) | 135 | 134
participants | 81 | 9
Statistical Analysis 1: Comparison: PEP005 (Ingenol Mebutate) Gel vs Vehicle Gel; Test type: Superiority or Other; p = 0.001, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Time Frame: 57 days
Description: For the safety population, the total sample size was 132 patients who received PEP005 Gel (2 patients never received study medication and one patient actually received vehicle gel) and 135 patients who received vehicle gel.
Arm/Group | PEP005 (Ingenol Mebutate) Gel, 0.015% | Vehicle
Serious Adverse Events (participants affected / at risk) | 2/132 | 2/135
Other Adverse Events (participants affected / at risk) | 39/132 | 3/135
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEP005 (Ingenol Mebutate) Gel, 0.015% (N=132) | Vehicle (N=135)
Campylobacter infection (Infections and infestations) | 1 (1) | 0 (0)
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) — Severe, Not related, Recovered
Meniscus Lesion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Lateral meniscus tear due to work injury, Severe, Not related, Recovered
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Vascular pseudoaneurysm (Vascular disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PEP005 (Ingenol Mebutate) Gel, 0.015% (N=132) | Vehicle (N=135)
APPLICATION SITE PAIN (Skin and subcutaneous tissue disorders) | 25 | 0
APPLICATION SITE PRURITUS (Skin and subcutaneous tissue disorders) | 14 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For US sites: The institution and investigator agree not to publish the results of this study without prior written consent of the Sponsor. As used herein, the term "publish" shall include oral presentations,written abstracts, written manuscripts, etc.